CLINICAL TRIAL: NCT01129492
Title: Low-Level Laser Therapy in Chronic Autoimmune Thyroiditis: Randomized, Placebo Controlled Clinical Trial
Brief Title: Low-Level Laser Therapy in Chronic Autoimmune Thyroiditis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Danilo Bianchini Höfling, University of São Paulo General Hospital - Radiology Departament
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPPesq 375/05
Record Dates: First submitted 2010-05-14; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2009-04

CONDITIONS: Autoimmune Thyroiditis
Keywords: Autoimmune Thyroiditis, Laser, Therapy, Thyroid, Ultrasound
MeSH Terms: conditions — Thyroiditis, Autoimmune; Thyroid Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Laser (Placebo Comparator): Ten applications of placebo were performed (twice a week) with the same method and Laser equipment, which has a placebo function available with a red ordinary light indistinguishable of the Laser light.
  Interventions: Device: Low-level Laser therapy
- Active Laser (Active Comparator): Ten applications of low-level Laser therapy (twice a week) were performed with a continuous wave diode laser device (830nm, beam area of 0.2827cm2), using the punctual method, continuous emission mode, output power of de 50 mW and fluence of 70J/cm2.
  Interventions: Device: Low-level Laser therapy

INTERVENTIONS:
Device: Low-level Laser therapy — A continuous wave (CW) diode laser device (830nm, infrared) with a beam area of 0.2827cm2 and using the punctual method, continuous emission mode, output power of de 50mW and fluence of 70J/cm2 (40 seconds at the point of application).
  Other Names: Low intensity Laser therapy; Low power Laser therapy

SUMMARY:
The purpose of this study is to evaluate whether low-level Laser therapy is effective in ameliorating the thyroid function of patients with hypothyroidism caused by chronic autoimmune thyroiditis.

DETAILED DESCRIPTION:
Chronic autoimmune thyroiditis (CAT) is the most common cause of hypothyroidism in iodine-replete areas. An autoimmune dysfunction causes humoral and cellular responses that lead progressively to thyroiditis. There is no effective therapy available that can change the natural history of CAT, which presents a high incidence of hypothyroidism and requires continuous treatment with levothyroxine (LT4).

Laser light can be valuable since the local and systemic actions of low-level laser therapy (LLLT) have been shown to be effective in treating autoimmune diseases, such as rheumatoid arthritis and Sjogren's syndrome. There is also evidence suggesting that LLLT can facilitate regeneration of various tissues and, in animal thyroids, can lead to improvement in microcirculation and increases in serum triiodothyronine (T3) and thyroxine (T4) levels. Since the LLLT is a non-invasive, cost-effective and painless procedure, the objective of this randomized clinical trial was to evaluate the effectiveness of LLLT in patients with hypothyroidism caused by chronic autoimmune thyroiditis, based on patients' thyroid function, their concentration of thyroid autoantibodies, and the parameters of their ultrasonography study.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with hypothyroidism induced by chronic autoimmune thyroiditis (CAT). The presence of hypothyroidism, laboratory measurements and ultrasonography criteria were applied to diagnose CAT.
* Significantly elevated concentrations of thyroid peroxidase (TPOAb) and/or thyroglobulin (TgAb) autoantibodies
* Ultrasonography results consistent with CAT
* Patients undergoing LT4 treatment
* Normal (or almost normal) levels of triiodothyronine (T3), thyroxine (T4), free T4 and thyrotropin (TSH)

Exclusion Criteria:

* Use of immunosuppressants, immunostimulants, or other drugs that could interfere with the production, metabolism and transport of thyroid hormones
* CAT with normal thyroid function
* CAT with subclinical hypothyroidism
* Thyroid nodules
* Hypothyroidism stemming from post-partum thyroiditis (up to 18 months after gestation)
* History of Graves' disease
* Thyrotropin receptor antibody (TRAb) detectable
* Prior treatment with radioiodine
* Tracheal stenosis
* Pregnancy
* History of ionizing irradiation and/or neoplasia in the cervical area
* Previous surgical intervention in the thyroid
* Thyroid hypoplasia
* Ectopic thyroid
* Serious illness (cancer, ischemic coronary artery disease, stroke, kidney or liver failure, etc.)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The main outcome measure was to gauge the effectiveness of applying LLLT in patients with hypothyroidism caused by CAT evaluated by a significant reduction of the levothyroxine (LT4) mean dose (µ/day) 9 months post-LT4 withdrawal. | LT4 dose, concentrations of T3, T4, free T4 and TSH were evaluated and compared before intervention and 9 months post-LT4 withdrawal.
  All patients enrolled in the study were undergoing LT4 treatment. They received 10 applications of LLLT or placebo. Thirty days after intervention, LT4 was discontinued in all patients and, if required, reintroduced. T3, T4, free T4 and TSH levels (all laboratory personnel was blinded), were assessed pre-LLLT and then 1, 2, 3, 6 and 9 months post-LT4 withdrawal. The LT4 mean dose pre-LLLT and 9 months post-LT4 withdrawal was compared both in face of normal levels of T3, T4, free T4 and TSH to evaluate LLLT effectiveness.

SECONDARY OUTCOMES:
Evaluate the LLLT efficacy in reducing thyroid autoantibodies concentrations. | Thyroid autoantibodies were determined and compared pre-intervention and 9 months post-LT4 withdrawal.
  Thyroid peroxidase (TPOAb) and thyroglobulin (TgAb) autoantibodies were both determined prior to LLLT and in the 1st, 2nd, 3rd, 6th and 9th months after LT4 withdrawal. All laboratory personnel was blinded to treatment assignment throughout the study.
Evaluate the LLLT efficacy by quantitative and qualitative ultrasonography parameters. | The ultrasonography parameters observed pre-LLLT were compared with those observed 30 days post-LLLT.
  B-mode sonography (volume, texture and echogenicity using computerized histogram) as well as power Doppler (vascularization) and pulsed Doppler (maximal systolic peak velocity and resistance index for the thyroid arteries) were performed and compared pre- and 30 days post-intervention by only one experienced and blind investigator, during the use of the same doses of LT4.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo B Höfling, Dr., Principal Investigator — University of São Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Hofling DB, Chavantes MC, Acencio MM, Cerri GG, Marui S, Yoshimura EM, Chammas MC. Effects of low-level laser therapy on the serum TGF-beta1 concentrations in individuals with autoimmune thyroiditis. Photomed Laser Surg. 2014 Aug;32(8):444-9. doi: 10.1089/pho.2014.3716. PMID 25101534